CLINICAL TRIAL: NCT05858749
Title: Clinical Effectiveness of First-Line Immuno-oncology (IO) Combination Treatment and Subsequent Lines of Therapy in Patients With Metastatic Renal Cell Carcinoma (mRCC) in the International Metastatic Renal Cell Carcinoma Database Consortium (IMDC)
Brief Title: A Study to Learn About the First and Later Lines of Medicines in Treating People With Metastatic Renal Cell Carcinoma (mRCC).
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061100
Record Dates: First submitted 2023-04-18; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Kidney cancer; Metastatic renal cell carcinoma (mRCC); International Metastatic Renal Cell Carcinoma Database Consortium (IMDC); Immunotherapy.
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with mRCC: Patients with mRCC in the IMDC

SUMMARY:
The purpose of this study is to learn about the effectiveness of the first and later lines of medicines on clinical outcomes in people with mRCC.

The study includes participants who:

* are 18 years old or above and have mRCC
* took medicines that use the bodies immunity to fight against cancer as their first choice of treatment
* took other medicines after taking the above first choice of treatment

This is a study that looks into the data collected through a particular database from selected academic clinical sites participating in this study. The data of interest include:

* the length of time between the start of a patient's treatment and the end of treatment
* the length of time between the start of treatment and death
* physician assessment of a patient's response to treatment

We will compare the experiences of people receiving different combinations of treatments and see if there are any differences in the effectiveness of these medicines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mRCC
* Age 18 years or over at the time of mRCC diagnosis
* Received IO combination treatment in 1L such as receiving ipilimumab + nivolumab or an axitinib-based regimen (ie, axitinib + pembrolizumab or axitinib + avelumab) as 1L
* Received subsequent treatments following 1L (e.g., 2L, 3L)
* Actively treated at an IMDC clinical center (to avoid incomplete data)

Exclusion Criteria:

- There are no exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective, longitudinal cohort study that involves the analysis of data collected through the IMDC database from selected academic clinical sites participating in this study.
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Demographical characteristics | From Time of Initiation of First-line (1L) Immuno-oncology (IO) combination therapy to death (up to 60 months)
  Gender Age at time of 1L initiation Race Region indicator (i.e., US vs. ex-US)
Date of mRCC diagnosis | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
Prior nephrectomy status | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
Date of nephrectomy (if applicable) | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
Tumor characteristics | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
  Histology type (i.e., clear cell vs. non-clear cell RCC) Number of metastatic sites (e.g., 1 site or more than 1 site) Site of metastases (e.g., brain, bone, lung)
IMDC risk score | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
  Assessed on index date and at initiation of each LOT
Number of lines of therapy received by each patient | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
Treatment agents received at each line of therapy | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
Duration of each line of therapy | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
Time from discontinuation of previous line of therapy to initiation of subsequent line of therapy | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
Reason for discontinuation for each line of therapy | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
Time to treatment discontinuation (TTD) | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
  Defined as the time from treatment initiation to discontinuation of each therapy due to any reason including progression, death, or toxicity
Time to next treatment (TTNT) | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
  Defined as time from the initiation of 1L treatment to initiation of subsequent therapy or death
Physician-assessed best response | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
  Overall best response rate (complete or partial) Stable disease Progressive disease
Overall survival | From Time of Initiation of 1L IO combination therapy to death (up to 60 months)
  Defined as the time between initiation of 1L IO combination therapy to death

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Headquarters, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4061100